CLINICAL TRIAL: NCT03302663
Title: The Value of Advanced Imaging Sequences for Fetal MRI in Clinical Practice
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Collaborators: University of Sheffield (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STH16555
Record Dates: First submitted 2017-06-20; First posted 2017-10-05 (Actual); Last update posted 2025-06-04 (Actual); Status verified 2025-05

CONDITIONS: Fetal Conditions
Keywords: Fetal bone heart abnormality
MeSH Terms: interventions — Magnetic Resonance Imaging

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to appropriate arm depending on outcome of routine obstetric screening
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Patients attending for a clinical scan (Other): Patients attending for a clinical scan will be offered 2-4 extra sequences. The additional sequences and compare them to the currently established ones.
  Interventions: Diagnostic Test: MRI scan
- Patients who have requested a TOP (Other): Women who have requested a termination of pregnancy (TOP) will be asked if they are willing to have a fetal MRI at 3T performed prior to the TOP. The images obtained will be compared to either images done clinically at 1.5T before the TOP request (if done and with the patients consent) or to images obtained at 1.5T of a similar gestation and pathology that the investigators obtained in a previous research study.
  Interventions: Diagnostic Test: MRI scan
- Patients with fetal heart abnormality (Other): The investigators plan to recruit patients with a fetus with heart abnormality on ultrasound and compare the MRI findings with the ultrasound findings and the clinical outcome.
  Interventions: Diagnostic Test: MRI scan
- Patient fetal bone abnormalities (Other): The investigators would like to ask women who have a fetus with bone abnormalities if they would be willing to have a fetal MRI. The findings will be compared to the ultrasound findings and the clinical or pathological findings after delivery.
  Interventions: Diagnostic Test: MRI scan

INTERVENTIONS:
Diagnostic Test: MRI scan — Addition of advanced imaging sequences for fetal MRI

SUMMARY:
This project is split into 4 sections:

1. Can improvements be made in the Magnetic resonance imaging sequences used to image the fetus in order to improve diagnostic accuracy?
2. Does 3T improve the quality and diagnostic value of fetal MRI when compared to 1.5T
3. Can fetal MRI be used to image the fetal heart?
4. Can fetal MRI be used to image the fetal Bones?

DETAILED DESCRIPTION:
Fetal MRI is rapidly expanding but the choice of sequences (the combination of variables that produce the image and determine whether a specific tissue is highlighted at the expense of other tissues e.g. some sequences highlight areas with a high water content, others highlight tissues with a high fat content) is limited. Additional sequences have the potential to improve the diagnostic accuracy but need to be developed and assessed before replacing the current choices. In addition it is not possible to continue to add sequences to the list used in clinical practice as each one takes time, which is limited in clinical practice. They may also allow other body areas to be imaged successfully e.g. bones and heart that are not currently imaged to a diagnostic level to be useful in clinical practice.

Until recently fetal MRI was restricted in the United Kingdom (UK) to magnet strengths of 1.5T although 3T was safely used in the rest of Europe. The restrictions have been lifted and 3T can now be used in the clinical setting for fetal MRI. The clinical value of this has not been established (1) In this pilot study the investigators will aim to answer the above 4 questions.

1. Currently the T2 SSFSE is used as the main sequence and in some institutions supplemented by T1 and diffusion-weighted imaging (DWI). The investigators wish to look at other sequences that may be better than these for imaging certain areas of the baby. The investigators have noted that the images used for imaging the placenta ( Balanced gradient echo) show the edges of tissues well but do not give much internal detail. However these images would be useful in cases of babies with cysts and may show the extension of the cyst more clearly than the T2. However it is not possible to simply add extra sequences to the scans as this takes extra time and is not appropriate in the clinical setting. This pilot study will allow evaluation of the sequences and formal comparison by a world-leading expert. This information will be used to guide local clinical practice but also with further development in the future to develop national guidelines.
2. 3T can now be used in the UK to image the fetus. Prior to imaging clinically at 3T it is necessary to establish if there is any additional benefit. This pilot will allow us to compare historical 1.5T images with 3T images to assess the potential benefit prior to a larger study.
3. Currently the fetal heart appears as a black ill-defined mass on the images. The investigators hope to use the balanced gradient echo sequence to image the heart. Initially the investigators would like to be able to image 4 chambers reliably and then to see if known pathology can be detected. If this is possible a larger study will be designed for further development. The question the investigators are asking is a very simple - can the investigators image the fetal heart? ' Yes/no and if so can the investigators reliably see 4 chambers? Yes/no. This will not need quantitative analysis.
4. Similar to 3 as currently no definition in fetal bone is seen. The investigators wish to apply sequences that reliably define the bone and then pilot these in cases with known bone pathology.

ELIGIBILITY:
Inclusion Criteria:

* Pregnant women who are attending the fetal medicine clinic and are asked to consider an MRI scan to provide information to help manage the current pregnancy.
* Pregnant women requesting a termination of pregnancy who will allow us to do fetal MRI at 3T prior to the termination.

Exclusion Criteria:

* Contraindication to MRI
* Severe claustrophobia

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Pregnant females
Enrollment: 150 (Estimated)
Dates: Start 2013-08-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Establish the value of advanced imaging sequences for fetal MRI in clinical practice | 3 years
  Part 1: improved imaging sequences that show areas better than the original sequences.
  Part 2: improved image quality when compared to similar (historical)cases done at 1.5T.
  Part 3 and 4: imaging of the fetal heart and bone that will be useful clinically (currently the images are not good enough to provide information for diagnosis and management)
  Overall improved image detail and quality to aid diagnosis and management.

CONTACTS AND LOCATIONS:
Overall Officials: Elspeth Whitby, Principal Investigator — University of Sheffield and Sheffield Teaching Hospitals NHS Foundation Trust
Locations (1):
- Sheffield Teaching Hospital NHS Foundation Trust, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided